CLINICAL TRIAL: NCT03603587
Title: Bioclinical Study of Scalp Photoaging of a Population Male Over 65 Years Old. Mono-centric Prospective Study
Brief Title: Bioclinical Study of Scalp Photoaging of a Population Male Over 65 Years Old.
Acronym: BACCHUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organisation issues
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18CH035; 2018-A00714-51 (Other: ANSM)
Record Dates: First submitted 2018-06-07; First posted 2018-07-27 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Skin Aging; Skin Cancer
Keywords: biologic markers; skin cancer; solar aging of skin; alopecic scalp
MeSH Terms: conditions — Skin Neoplasms | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a prospective mono-centric study of the physiopathology of cutaneous aging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who will benefit from the removal of a scalp tumour (Experimental): Patients who will benefit from the removal of a scalp tumour in the alopecic zone will be recruited in the dermatology department of the St-Etienne University Hospital.
  They will have biopsy, blood sample, examination of the scalp, questionnaire on sun exposure, Norwood scale, scinexa score, questionnaire of clinicals signs and questionnaire of the history of the hair loss.
  Interventions: Procedure: biopsy; Diagnostic Test: blood sample; Diagnostic Test: questionnaire on sun exposure; Diagnostic Test: examination of the scalp; Diagnostic Test: Norwood scale; Diagnostic Test: questionnaire of clinicals signs; Diagnostic Test: scinexa score; Diagnostic Test: questionnaire of the history of the hair loss

INTERVENTIONS:
Procedure: biopsy — Biopsy 4 to 5 mm from the distal part of the tips of the excision pieces. Three biopsies of 3 mm, made with punch, occipital hair zone (ZT) A completely painless sample, using a swab (soaked with a buffer solution) on the scalp of the ZH and ZT zone.
Diagnostic Test: blood sample — Blood sample will be collected for performed for HIV serology, B and C hepatitis.
Diagnostic Test: questionnaire on sun exposure — Questionnaire on sun exposure will be completed by patients.
Diagnostic Test: examination of the scalp — A complete examination of the scalp will be completed by dermatologist.
Diagnostic Test: Norwood scale — Norwood scale measure the evolution of baldness. It will be completed by dermatologist.
Diagnostic Test: questionnaire of clinicals signs — Questionnaire of clinicals signs will be completed by dermatologist and patient.
Diagnostic Test: scinexa score — It's a assessment score of skin aging. It will be completed by dermatologist.
Diagnostic Test: questionnaire of the history of the hair loss — Questionnaire of the history of the hair loss will be completed by dermatologist and patient.

SUMMARY:
The aging of skin, especially that of the scalp, is a combination of intrinsic and extrinsic aging factors secondary to the chronic sun exposure. For men with an alopecia genetic (= bald men), the solar part, in skin aging process, is major.

The helio-dermal scalp is frequently the site of cancers mainly after 65 years. Objectives are to identify specific biomarkers involved in the photo-aging of the alopecic scalp

DETAILED DESCRIPTION:
Investigators can also hope to understand and to explain the inter-individual inequality of the aging of skin. They can hope to a better understanding of the biological mechanisms between photo-induced skin aging and photo-induced carcinogenesis.

Investigators propose to study 40 male patients aged 65 and over in order to compare the state of aging of their scalp skin in the alopecic zone :

not hairy photo-exposed (= ZH sun damage zone) versus occipital hair zone protected photo (= ZT control zone).

Patients will be recruited in the dermatology department of the St-Etienne University Hospital who will benefit from the removal of a scalp tumour in the alopecic zone.

This study aims to identify biological markers, by transcriptomic analysis, associated with aging of the scalp, by comparing for each patient the skin of the scalp exposed to the light ("ZH") to an unexposed witness skin ("ZT").

The study will include :

* examinations to characterize components of the scalp: transcriptomic, proteomic and immunohistochemical analysis of skin biopsies, and a swab sampling will identify the cutaneous microflora of the scalp
* noninvasive examinations, in vivo

ELIGIBILITY:
Inclusion Criteria:

* Requiring excision of an alopecic scalp lesion
* from consent signed
* Patient affiliated or entitled to a social security.

Exclusion Criteria:

* scalp infection
* inflammatory disease of the scalp
* genetic disease with even partial expression of the scalp
* medical treatment of scalp less than 3 weeks old
* antecedent radiotherapy of the cephalic extremity
* prior surgery of the scalp with regard to the area sampled
* Application of hair implants, or any other surgical or medical procedures of the scalp
* Washing of the scalp or application of a cosmetic product for less than 48 hours
* Artificial hair coloring.
* any contraindication to surgical excision

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — - Men
Enrollment: 1 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Scalp skin biomarkers | at the surgery (about 28 days after the inclusion)
  Comparison of scalp skin biomarkers. It's compare cell differentiation, cell proliferation, cellular pigmentation, cell adhesion, cytoskeleton, aging and cellular senescence, extracellular matrix, antioxidant activity and inflammation.

SECONDARY OUTCOMES:
Differential expression profile of proteomic biomarkers | 28 days
  The profile will be evaluated by relative quantification results of proteomic analyzes by a Shot-Gun Label-Free strategy.
Data of thickness measurements of the 3 layers of the skin | 28 days
  Data will be examined by OCT examination (Optical Coherent Tomography): measuring the intensity of the dermis shine and the thickness of the epidermis.
scalp microflora | 28 days
  Microflora will be evaluated by high-throughput sequencing (Illumina MiSeq) of the V1-V3 region of the ribosomal RNA (bacteria) and Internal Transcribed Spacer 1 (eukaryotes: yeasts) and evaluation of the amount of P. acnes of the scalp by quantitative RT-PCR of the lipase A gene.
Percentage of anisotropy of the tensile forces of the skin | 28 days
  This percentage will be evaluated by silicone casts
histology | 28 days
  Skin aging is evaluated by histological examination: optical and biophotonic microscopy, semi-quantitative measurements of extracellular matrix markers such as collagens and elastin.
Heterogeneity of pigmentation | 28 days
  Heterogeneity of pigmentation will be measured using a numerical index (0 to 100) of heterogeneity, using data from dermatoscopic images.
Scinexa score (SCore for INtrinsic and EXtrinsic skin Aging) | 28 days
  The aging of the skin is evaluated by a semi-quantitative composite of 23 clinical variables : the scinexa score The global SCINEXA score (from 0 to 69. 0 = no skin aging and 69 = severe skin aging ) was obtained by adding the scores of each variable from 0 to 3.
  0 = none, 1 = mild, 2 = moderate and 3 = severe.
The measurement of the thickness of the dermis | 28 days
  ultrasound examination: measurement in mm of the thickness of the dermis and the hypodermis
The measurement of the morphology of the dermal junction epidermis | 28 days
  examination in MCIV: measurement of the morphology of the dermal junction epidermis by semi-quantitative in vivo confocal microscopy
Solar exposure score | 28 days
  Solar exposure score : to assess in different periods
  1. period of 10 to 17 years old
  2. period of 18 to 40 years old
  3. period of 41 to 60 years old
  4. period since 61 years old
  Each period contains same questions. Each item being rated in 5 answer choice from 1 to 5 (never, rarely, sometimes, often or very often) and two questions concern the zone where the patient live.
Norwood's scale | 28 days
  The Norwood Scale is a set of images that depict the different stages of male pattern hair loss.
  The Norwood scale is composed of 12 images. Each image corresponds to one level. There is 7 levels (I , II, II A, III, III vertex, III A, IV, IVA, V, VA, VI, VII) Type I. Minimal hair loss. Type VII. The most severe form of hair loss. Little hair on the front or top of the head.

CONTACTS AND LOCATIONS:
Overall Officials: JEAN LUC PERROT, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zouboulis CC, Makrantonaki E. Clinical aspects and molecular diagnostics of skin aging. Clin Dermatol. 2011 Jan-Feb;29(1):3-14. doi: 10.1016/j.clindermatol.2010.07.001. PMID 21146726
- [Background] Uitto J. Understanding premature skin aging. N Engl J Med. 1997 Nov 13;337(20):1463-5. doi: 10.1056/NEJM199711133372011. No abstract available. PMID 9358147
- [Background] Shin MH, Rhie GE, Park CH, Kim KH, Cho KH, Eun HC, Chung JH. Modulation of collagen metabolism by the topical application of dehydroepiandrosterone to human skin. J Invest Dermatol. 2005 Feb;124(2):315-23. doi: 10.1111/j.0022-202X.2004.23588.x. PMID 15675949
- [Background] Rock K, Grandoch M, Majora M, Krutmann J, Fischer JW. Collagen fragments inhibit hyaluronan synthesis in skin fibroblasts in response to ultraviolet B (UVB): new insights into mechanisms of matrix remodeling. J Biol Chem. 2011 May 20;286(20):18268-76. doi: 10.1074/jbc.M110.201665. Epub 2011 Mar 17. PMID 21454612
- [Background] Varani J, Spearman D, Perone P, Fligiel SE, Datta SC, Wang ZQ, Shao Y, Kang S, Fisher GJ, Voorhees JJ. Inhibition of type I procollagen synthesis by damaged collagen in photoaged skin and by collagenase-degraded collagen in vitro. Am J Pathol. 2001 Mar;158(3):931-42. doi: 10.1016/S0002-9440(10)64040-0. PMID 11238041